CLINICAL TRIAL: NCT00809952
Title: Ultrasound Guided Artificial Insemination
Acronym: UGAI
Status: Completed | Type: Observational
Sponsor: Hospital de Cruces (Other)
Other Study IDs: HUMREP-08-0656
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2008-12-17 (Estimated); Status verified 2008-12

CONDITIONS: Insemination

GROUPS / COHORTS (1):
- Recombinat FSH
  Interventions: Procedure: recombinant FSH

INTERVENTIONS:
Procedure: recombinant FSH

SUMMARY:
The purpose of this study is to ascertain whether using ultrasound guidance during intrauterine insemination (IUI) could increase pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* The woman's inclusion criteria in our IUI program were at least one patent tube, normal cavity, basal FSH < 10 mU/mL and age under 40 years.
* IUI with husband's sperm (IUI-H) was indicated when, after sperm preparation, at least 5 million motile spermatozoa were recovered; this was performed in 58 cases (79.45%).
* In the remaining 15 cases (20.55%), IUI was performed with donor sperm (IUI-D) either because of azoospermia (n=6) failure to recover spermatozoa during testicular biopsy (n=5) or in women without a male partner (n=4).

Exclusion Criteria:

* Previous infertility treatments had been carried out.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Human Reproduction Unit, Cruces-Baracaldo, Basque Country, Spain

REFERENCES:
- [Derived] Ramon O, Matorras R, Corcostegui B, Meabe A, Burgos J, Exposito A, Crisol L. Ultrasound-guided artificial insemination: a randomized controlled trial. Hum Reprod. 2009 May;24(5):1080-4. doi: 10.1093/humrep/den498. Epub 2009 Feb 5. PMID 19196748